CLINICAL TRIAL: NCT03180398
Title: Pilot Study of Using Multi-parametric Magnetic Resonance Imaging for Organ Delineation and Tumor Response Assessment of Prostate Cancer Patients Being Treated With Radiation Therapy
Brief Title: Multi-parametric Magnetic Resonance Imaging for Prostate Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Stephen Brown, Director, Radiobiology Research Laboratories, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prostate Imaging 10911
Record Dates: First submitted 2017-06-05; First posted 2017-06-08 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Multi-parametric MRI for Prostate Cancer (Experimental): MRI will be acquired for prostate cancer patients undergoing radiation treatment.
  Interventions: Device: Multiparametric MRI

INTERVENTIONS:
Device: Multiparametric MRI — MRI will be acquired before, during and after radiation treatment to evaluate treatment response

SUMMARY:
This is a pilot study of implement multi-parametric MR imaging for organ delineation and tumor response assessment of prostate cancer patients being treated with radiation therapy.

DETAILED DESCRIPTION:
The study aims to generate intraprostatic lesions maps based on imaging, perform the treatment planning to compute the highest feasible simultaneous boosting dose to intraprostatic lesion and characterize longitudinal changes in imaging characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma

Exclusion Criteria:

* Patients with metal fragments or implanted devices such as pacemakers and aneurysm clips are not eligible for the study considering

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multi-parametric MRI for Prostate Cancer
Started | 9
Completed | 9 (Study closed due to lack of accrual.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Multi-parametric MRI for Prostate Cancer
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Detection of Imaging Biomarkers to Localize the Intraprostatic Lesions and Predict Radiation Treatment Response
Description: Identify the radiomics features selected from multimodal MRI to distinguish the dominant lesions from the normal tissues within the prostate. Track the changes of these features with longitudinal MRI scans to identify its correlation with the local control.
Time Frame: 2 years
Population: Radiomics requires sufficient patient number. Not enough patients were included for radiomics analyses.
  PI left institution and country. The data was not collected so analysis could not be completed.
Groups:
- Multi-parametric MRI for Prostate Cancer: MRI were to be acquired for prostate cancer patients undergoing radiation treatment.
  Multiparametric MRI: MRI was to be acquired before, during and after radiation treatment to compare with treatment response.
  The Principal Investigator (Ning Winston Wen) departed the institution, accrual was low and the study was closed.
Arm/Group | Multi-parametric MRI for Prostate Cancer
Number analyzed (Participants) | 0
Statistical Analysis 1: Comparison: Multi-parametric MRI for Prostate Cancer; Test type: Superiority — It was hoped to compare radiomics features, using non-parametric tests, but this was not possible because of the small number of patients accrued; Not enough patients were accrued for radiomics analysis. PI left institution and country. Analysis could not be completed

2. Primary Outcome: Tumor Response
Description: Tumor response as measured by an increase in PSA.
Time Frame: 2 years
Population: The patient number was too small for the planned radiomics analysis. The study was closed. The data was not collected so analysis could not be completed.
  PI left institution and country. Analysis could not be completed.
Groups:
- Multi-parametric MRI for Prostate Cancer: MRI will be acquired for prostate cancer patients undergoing radiation treatment.
  Multiparametric MRI: MRI will be acquired before, during and after radiation treatment to evaluate treatment response
  The Principal Investigator (Ning Winston Wen) left the institution. Accrual was slow and low. The study was closed.
Arm/Group | Multi-parametric MRI for Prostate Cancer
Number analyzed (Participants) | 0
Statistical Analysis 1: Comparison: Multi-parametric MRI for Prostate Cancer; Test type: Other — Analysis could not be completed; PI left institution and country. Analysis could not be completed

ADVERSE EVENTS:
Time Frame: 2 years
Description: Only images of patients were acquired. There is no risk to the patients.
Arm/Group | Multi-parametric MRI for Prostate Cancer
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03180398/Prot_002.pdf
  • Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT03180398/SAP_004.pdf
  • Informed Consent Form (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT03180398/ICF_001.pdf